CLINICAL TRIAL: NCT05176379
Title: Endothelial Derived Hyperpolarization Factor and Regulation of Cerebral and Muscle Blood Flow
Brief Title: Endothelial Derived Hyperpolarization Factor and Vascular Control
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 14056
Record Dates: First submitted 2021-12-01; First posted 2022-01-04 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Healthy
Keywords: brain blood flow; muscle blood flow; endothelial function
MeSH Terms: interventions — Fluconazole

STUDY DESIGN:
Intervention Model Description: Randomized, single-blind, Placebo controlled, crossover design
Who Masked: Participant
Masking Description: Participants will receive a placebo instead of fluconazole
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- fluconazole (Experimental): fluconazole tablet/pill 150 mg, single acute dose
  Interventions: Drug: Fluconazole 150 mg
- Placebo (Placebo Comparator): 250 mg pill microcrystalline Cellulose, single acute dose
  Interventions: Drug: Fluconazole 150 mg

INTERVENTIONS:
Drug: Fluconazole 150 mg — A single acute 150 mg dose
  Other Names: placebo

SUMMARY:
Most cardiometabolic diseases are characterized by increased muscle sympathetic nerve activity (MSNA) during rest and exercise which contributes to poor health outcomes. In healthy humans during muscle contraction, there is a blunting of skeletal muscle vascular responsiveness to increases in MSNA. However, the exact mechanisms involved are unknown although, best evidence suggests that the mechanism is endothelium derived, but nitric oxide (NO) and prostaglandin (PG) independent. Endothelium-derived hyperpolarizing factor (EDHF) is a NO and PG independent vasodilator in both cerebral and skeletal muscle circulations, however, it is unknown if EDHF contributes to vascular responsiveness during elevated MSNA. The application of lower body negative pressure (LBNP) is a safe and non-invasive manipulation that can be used to increase MSNA causing vasoconstriction in humans. Therefore, the purpose of this experiment is to determine if acute inhibition of EDHF alters central and peripheral vascular responses to LBNP at rest and during dynamic exercise. Thereby, providing evidence by which EDHF contributes to vascular control in healthy humans and identify it's potential as a therapeutic target for cardiometabolic diseases that are characterized by elevated MSNA

DETAILED DESCRIPTION:
The purpose of this study is to investigate the importance of the endothelium-derived hyperpolarizing factor (EDHF) in regulation of muscle and brain blood flow during rest, sympathetic activation via lower body negative pressure (LBNP), and during rhythmic exercise. We hypothesize that acute inhibition of EDHF will blunt cardiovascular responses and decrease peripheral tissue oxygenation (specifically in the brain and muscle) in response to LBNP during rest and during exercise. This work will provide evidence that EDHF counter acts sympathetic nervous activity in healthy humans, thereby highlighting EDHF as a potentially crucial mechanism in human vascular control. Ultimately this work will provide basic knowledge need to open longer treatment windows and potentially novel therapies for cardiovascular complications from cardiometabolic diseases.

To test these hypotheses, we will complete two specific aims:

I) To test the hypothesis whether EDHF inhibition alters sympathetic restraint muscle vasculature (termed, sympatholysis), we will compare changes in oxygenated hemoglobin (O2Hb), deoxygenated hemoglobin (HHb), Cardiac Output (CO) and Mean Arterial Pressure (MAP), Total Peripheral Resistance (TPR), Tissue Oxygen Saturation Index (TSI) during sympathetic activation (LBNP) and Handgrip exercise in two conditions: placebo vs. acute EDHF inhibition (Fluconazole).

II) To test the hypothesis whether EDHF inhibition alters regulation of cerebral blood flow during rest and sympathetic activation (LBNP), we will compare changes in cerebral vascular conductance index (CVCi), cerebral TSI as well as gain, coherence, and phase in transfer functional analysis during the exposure to Lower Body Negative Pressure (LBNP) in two conditions: placebo vs. acute EDHF inhibition (Fluconazole)

ELIGIBILITY:
Inclusion Criteria:

* Normotensive (systolic blood pressure < 130 mmHg and/or diastolic blood pressure < 85 mmHg) individuals
* Individuals free of cardiovascular disease and metabolic disease
* Individuals free of any form of autonomic dysfunction
* Individuals with a BMI under 30 kg/m²
* Women that are premenopausal with a regular menstrual cycle (26-30 days)

Exclusion Criteria:

* Smokers, tobacco users (regular use in the last 6 months)
* Individuals with a blood pressure greater than 130/85
* Subjects who use Amiodarone, Sulphaphenazole
* Subjects who use S-warfarin, Tolbutamine, Phenytoin, Lonafarnib
* Cardiometabolic medication use (e.g. anti-hypertensives, insulin-sensitizing, statins)
* Sex hormone replacement medical use (e.g. testosterone, estrogen, progesterone)
* Pregnancy

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-02-19 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Near-Infrared Spectroscopy | up to 4 hours
  Concentrations of Oxygen, deoxy, and Total Hemoglobin (micro molar)
Transcranial Doppler Ultrasound | up to 4 hours
  middle cerebral artery blood velocity

SECONDARY OUTCOMES:
Wireless electrocardiogram | up to 4 hours
  heart rate
Finger photoplethysmography | up to 4 hours
  Mean Arterial Pressure

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy M Kellawan, PhD, Principal Investigator — University of Oklahoma
Locations (1):
- Department of Health and Exercise Science, Norman, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual participant data